CLINICAL TRIAL: NCT02644096
Title: Rehabilitation of Patients Aged 65 and Over After Total Hip Replacement - Based on Patients´Health Status
Brief Title: Rehabilitation of Patients After THR - Based on Patients´Selfrated Health
Acronym: Rehab-THR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Sygekassernes Helsefond (Other); TrygFonden, Denmark (Industry); Region Zealand (Other)
Responsible Party: Principal Investigator, Britta Hørdam, Senior researcher, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Rehabilitation after THR
Record Dates: First submitted 2015-08-03; First posted 2015-12-31 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-07

CONDITIONS: Total Hip Replacement
Keywords: Rehabilitation; RCT; User Involvement; Self-Rated Health
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional treatment (No Intervention): After surgery, patients with total hip replacement are only seen once 3 months after surgery, and they have no further contact with the hospital.
- Intervention (Other): counselling and support after discharge from hospital
  Interventions: Other: counselling and support after discharge from hospital

INTERVENTIONS:
Other: counselling and support after discharge from hospital — patients were contacted by telephone 2 times after discharge from surgery by a specialist nurse, who followed an interview guide due to nursing-rehabilitation after THR
  Arms: Intervention

SUMMARY:
Objective: The investigators hypothesized that all areas of health status after total hip replacement could be improved in patients aged over 65 years and over by using telephone support and counselling 2 and 10 weeks after surgery compared with a control group receiving conventional care and treatment.

Design: A randomised clinical trial focusing on patients' health status by using SF-36 at 4 weeks pre- and 3 and 9 months postoperatively was carried out. Sample: 180 patients aged 65 and over were randomised 4 weeks preoperatively to either control or intervention groups. Measurements: Both groups received conventional surgical treatment, but the intervention group was interviewed by telephone 2 and 10 weeks after surgery. Patients were given counselling within eight main dimensions with reference to their postoperative situation.

Key-words: THR - elderly patients - health status - postoperative support - counselling

DETAILED DESCRIPTION:
Primary outcome: the physical dimensions in health status. The intervention could lead to an improvement of 50% in the physical health score on the SF-36 questionnaire.

Theoretical frame of reference: the nursing intervention in this study was based on the Murray and Maslow's theories of motivation combined with Piaget's theory of development in which the main goal is to promote and maintain patients' active involvement in their own care.

Intervention: All patients received the standard postoperative procedure in the hospital, which means discharge after 5-7 days and a clinical control in the outpatient department after 3 months. But the intervention group also received telephone support and counselling 2 and 10 weeks after surgery. The intervention was performed by the same nurse using a structured interview guide to identify the patients' perceptions of their current situations and need for further support and counselling of importance to their health status. Together the patients and the nurse assessed the patients' situation and areas of improvements. The assessment focused on eight main dimensions referring to the patients' situation after Total Hip Replacement (THR). (1) Wellbeing. (2) Expectations as to PF after surgery. (3) Expectations as to PF compared with those before surgery. (4) Symptoms (pain, leg-oedema, vertigo, sleep disturbance, nausea and other concerns) and (5) Problems with eating and appetite. (6) Fluid intake. (7) Ability to follow prescribed activity and exercise. (8) Need of support from family. For each of the problems identified,individual solutions were suggested and practical counselling was given by the investigator.

Statistical analysis: Data were processed by using the statistical program Statistical Package for Social Sciences (SPSS) version 13.0 (Boston, MA, USA). Ratio-scaled data from both groups (intervention and control) were compared by using parametric methods if data were normally distributed, but if not, nonparametric methods were used. Nominal scaled data were compared by using the chi-square test or using 95% CI around the association measure.

Categorical variables were compared using Pearson's chi-square test if appropriate. For continuous data, changes within the groups were analysed by using a paired t-test. Groups were compared using an unpaired t-test (for normally distributed data). p < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled to THR
* Being able to read and understand Danish

Exclusion Criteria:

* Patients not being able to participate or refused
* Any condition that makes the subject unable to participate in the opinion of the investigator.

Ages: 65 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 175 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2013-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out in two orthopaedic departments in Aarhus university hospital in Denmark in the period from January 2005 until May 2007. All patients were recruited from the hospitals waiting list.
Pre-assignment Details: 180 patients were given the SF-36 questionnaire preoperatively. 175 questionnaires were returned and so 175 patients were randomised into the study.
Period: Overall Study
Arm/Group | Conventional Treatment | Intervention
Started | 93 | 82
2 Week Interview | 0 (Not done in control group) | 68
10 Week Interview | 0 (Not done in control group) | 59
12 Week SF-36 Questionnaire | 68 | 59
9 Month SF-36 Questionnaire | 65 | 57
Completed | 65 | 57
Not Completed | 28 | 25
Not completed — Withdrawal by Subject | 28 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Treatment | Intervention | Total
Number analyzed (Participants) | 93 | 68 | 161
Age, Categorical [Count of Participants; unit: Participants] — The baseline information was collected from hospital records.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 93 | 68 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (8.1) | 75 (8.6) | 74.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 33 | 78
  Male | 48 | 35 | 83
Region of Enrollment [Number; unit: participants]
  Denmark | 93 | 68 | 161

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Dimensions in Health Status of Elderly Patients From 4 Weeks Pre Operatively to 9 Months Post Operatively After THR. Health Status is Measured by the Questionnaire Short-form 36 (SF-36).
Description: The health status was assessed by Short-Form 36 (SF-36) which is a self-administered generic questionnaire that has been shown to be reliable and valid for measuring functioning, well-being and general health status. The instrument measures the eight health dimensions listed in figure 3. Reflecting the impact of both dysfunctions and general health perception the questionnaire measures: physical function (PF), role physical (RF), bodily pain (BP), social function (SF) role emotional (RE), general health (GH), vitality (VT) and mental health (MH). The questions related to each dimension are scored on a scale from 0 (worst score) to 100 (best score).
  All patients who had been consecutively admitted for THR were mailed an introduction letter together with a questionnaire containing a number and a prepaid return envelope. In the questionnaire they were asked to give demographic data and assess their health status
Time Frame: Four weeks preoperatively and nine moths after discharge.
Population: Patients who have completed the study and contributed with answers on the SF-36 questionnaire.
Measure: Mean (95% Confidence Interval); unit: Scores on SF-36 questionnaires
Groups:
- Intervention: counselling and support after discharge from hospital
  counselling and support after discharge from hospital: patients were contacted by telephone 2 times after discharge from surgery by a specialist nurse, who followed an interview guide due to nursing-rehabilitation.after THR.
Arm/Group | Conventional Treatment | Intervention
Number analyzed (Participants) | 65 | 57
Scores on SF-36 questionnaires
  Changes in physical function after 3 months | 9.6 [4.4 to 14.7] | 17.8 [12.4 to 23.1]
  Changes in general health after 3 months | 1.2 [-4.8 to 2.5] | 7.3 [3.4 to 11.1]
  Changes in mental Health after 3 months | 4.2 [0.4 to 8.8] | 11.1 [5.9 to 16.3]
  Changes in physical health after 9 months | 16.9 [10.3 to 23.6] | 17.9 [11.9 to 23.9]
  Changes in general health after 9 months | 1.4 [-7.4 to 4.5] | 5.7 [1.6 to 9.9]
  Changes in mental health after 9 months | 8.4 [3.1 to 13.7] | 12.1 [5.8 to 18.4]
Statistical Analysis 1: Comparison: Conventional Treatment vs Intervention; Power calculation in this study was based on findings in a previous cross-sectional study. The physical dimensions in health status was the primary outcome variable. The mean physical score was 49.4, SD was 26.1; alpha in this study was set to 5% and β to 20%. We considered that the intervention could lead to an improvement of 50% in the physical health score and were willing to overlook a difference in score of 12. When the sample size was calculated, 68 patients were needed in both groups; Test type: Superiority or Other; p < 0.05, unpaired t-test — Changes in physical function after 3 months

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Conventional Treatment | Intervention
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/68
Other Adverse Events (participants affected / at risk) | 0/93 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes